CLINICAL TRIAL: NCT02843022
Title: Enhancing Follow-up Mechanisms for Women at Risk for Postpartum Depression
Brief Title: Effectiveness of a Web-based Nursing Intervention in the Reduction of Postpartum Depression and Parenting Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Anselm College (Other)
Collaborators: Catholic Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NURS2015-3
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Depression, Postpartum
Keywords: postpartum; nursing; follow-up
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Active Comparator): Participant will receive the usual care provided by the nursing staff at Catholic Medical Center. A lactation consultant or childbirth educator attempts to call each patient within 2-3 weeks prior to discharge. Only one call is made, and a message left if the patient would like to call back.
  Interventions: Behavioral: Staff nurse phone follow-up
- Message Only (Experimental): Participant will receive the usual care, and in addition, will receive four standardized electronic messages weekly for six months postpartum. These will be one-way messages without the option to respond.
  Interventions: Behavioral: standardized electronic messages; Behavioral: Staff nurse phone follow-up
- Message and Nurse (Experimental): Participant will receive the usual care as well as the four standardized electronic messages/week for 6 months. Two of these weekly messages will be two-way, providing the option for the participant to respond "yes" to an offer to have a nurse call them. A nurse phone call if requested will be provided with a week.
  Interventions: Behavioral: standardized electronic messages; Behavioral: nurse phone call if requested; Behavioral: Staff nurse phone follow-up

INTERVENTIONS:
Behavioral: standardized electronic messages — supportive and educational short messages
  Other Names: text messages; email messages
  Arms: Message Only; Message and Nurse
Behavioral: nurse phone call if requested — If participant responds "yes" to an offer for a phone call, a nurse calls them within a week of this response
  Arms: Message and Nurse
Behavioral: Staff nurse phone follow-up — Usual care: hospital nurse or lactation consultant calls patient within 2-3 weeks prior to discharge. Message left if patient is not reached.

SUMMARY:
The purpose of the study is to determine whether a web-based nursing intervention delivered during the postpartum period will decrease symptoms of postpartum depression and parenting stress.

DETAILED DESCRIPTION:
The purpose of this randomized, controlled trial is to determine whether receiving standardized messages (text or email) from a postpartum nurse four times/week for 6 months after delivery will decrease symptoms of postpartum depression and parenting stress. Enrolled women will be randomized to one of three groups. The first group will receive the usual care, which is a phone call from a nurse within the first few weeks postpartum. The second group will receive four standardized messages each week, the content of which will include infant care, maternal self-care and inspirational material. The third group will receive the same four standardized messages each week, and in addition, two of these weekly messages will offer the option to respond with a request for a nurse to call them. Baseline data will be collected during the postpartum hospitalization, and follow-up will occur by email at 3 weeks, 3 months and 6 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Able to speak and read English
2. Access to a device which can receive text or email messages

Exclusion Criteria:

1. Non-English speaking,
2. No access to a device which can receive text or email messages
3. Age younger than 18 -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2015-11; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
postpartum depression symptoms | 6 months postpartum
  Measured by scores on the Edinburgh Postnatal Depression Scale (EPDS) at three time points

SECONDARY OUTCOMES:
breastfeeding outcomes | 6 months postpartum
  Duration and pattern of infant feeding
patient satisfaction/experience | 6 months postpartum
  Participant response to the experience of receiving messages and having the option to talk to a nurse (group 3), as well as their sense of connection to the hospital where they gave birth
Parenting stress | 6 months postpartum
  Scores on the Parenting Stress Index (PSI-4)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E. McCarter, PhD, RN, Principal Investigator — Saint Anselm College
Locations (1):
- Catholic Medical Center, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segre LS, O'Hara MW, Arndt S, Beck CT. Screening and counseling for postpartum depression by nurses: the women's views. MCN Am J Matern Child Nurs. 2010 Sep-Oct;35(5):280-5. doi: 10.1097/NMC.0b013e3181e62679. PMID 20706098
- [Background] Piette JD, Schillinger D. Applying interactive health technologies for vulnerable populations. In: King TE, Wheeler MB, eds. Medical management of vulnerable and underserved patients: Principles, practice and populations. New York: McGraw-Hill; 2007.
- [Background] Mood and Anxiety Disorders in Pregnant and Postpartum Women. J Obstet Gynecol Neonatal Nurs. 2015 Sep-Oct;44(5):687-9. doi: 10.1111/1552-6909.12734. Epub 2015 Jun 30. No abstract available. PMID 26126933
- [Background] Segre LS, O'Hara MW, Arndt S, Stuart S. The prevalence of postpartum depression: the relative significance of three social status indices. Soc Psychiatry Psychiatr Epidemiol. 2007 Apr;42(4):316-21. doi: 10.1007/s00127-007-0168-1. Epub 2007 Feb 13. PMID 17370048
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Earls MF; Committee on Psychosocial Aspects of Child and Family Health American Academy of Pediatrics. Incorporating recognition and management of perinatal and postpartum depression into pediatric practice. Pediatrics. 2010 Nov;126(5):1032-9. doi: 10.1542/peds.2010-2348. Epub 2010 Oct 25. PMID 20974776
- [Background] Knitzer J, Theberge S, Johnson K. Reducing maternal depression and its impact on young children: Toward a responsive early childhood policy framework. Project Thrive 2008.
- [Background] Paulson JF, Dauber S, Leiferman JA. Individual and combined effects of postpartum depression in mothers and fathers on parenting behavior. Pediatrics. 2006 Aug;118(2):659-68. doi: 10.1542/peds.2005-2948. PMID 16882821
- [Background] McLennan JD, Kotelchuck M. Parental prevention practices for young children in the context of maternal depression. Pediatrics. 2000 May;105(5):1090-5. doi: 10.1542/peds.105.5.1090. PMID 10790467
- [Background] Sills MR, Shetterly S, Xu S, Magid D, Kempe A. Association between parental depression and children's health care use. Pediatrics. 2007 Apr;119(4):e829-36. doi: 10.1542/peds.2006-2399. PMID 17403826
- [Background] Beck A, Crain AL, Solberg LI, Unutzer J, Glasgow RE, Maciosek MV, Whitebird R. Severity of depression and magnitude of productivity loss. Ann Fam Med. 2011 Jul-Aug;9(4):305-11. doi: 10.1370/afm.1260. PMID 21747101
- [Background] Brealey SD, Hewitt C, Green JM, Morrell J, Gilbody S. Screening for postnatal depression -- is it acceptable to women and healthcare professionals? A systematic review and meta-synthesis. Journal of Reproductive & Infant Psychology. 2010;28:328-344.
- [Background] Gjerdingen DK, Yawn BP. Postpartum depression screening: importance, methods, barriers, and recommendations for practice. J Am Board Fam Med. 2007 May-Jun;20(3):280-8. doi: 10.3122/jabfm.2007.03.060171. PMID 17478661
- [Background] McCarter-Spaulding D, Shea S. Effectiveness of Discharge Education on Postpartum Depression. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):168-72. doi: 10.1097/NMC.0000000000000236. PMID 27128643
- [Background] Furber G, Jones GM, Healey D, Bidargaddi N. A comparison between phone-based psychotherapy with and without text messaging support in between sessions for crisis patients. J Med Internet Res. 2014 Oct 8;16(10):e219. doi: 10.2196/jmir.3096. PMID 25295667
- [Background] Aguilera A, Munoz RF. Text Messaging as an Adjunct to CBT in Low-Income Populations: A Usability and Feasibility Pilot Study. Prof Psychol Res Pr. 2011 Dec 1;42(6):472-478. doi: 10.1037/a0025499. PMID 25525292
- [Background] Aguilera A, Berridge C. Qualitative feedback from a text messaging intervention for depression: benefits, drawbacks, and cultural differences. JMIR Mhealth Uhealth. 2014 Nov 5;2(4):e46. doi: 10.2196/mhealth.3660. PMID 25373390
- [Background] Le HN, Perry DF, Sheng X. Using the internet to screen for postpartum depression. Matern Child Health J. 2009 Mar;13(2):213-21. doi: 10.1007/s10995-008-0322-8. Epub 2008 Feb 16. PMID 18278545
- [Background] Drake E, Howard E, Kinsey E. Online screening and referral for postpartum depression: an exploratory study. Community Ment Health J. 2014 Apr;50(3):305-11. doi: 10.1007/s10597-012-9573-3. Epub 2013 Jan 3. PMID 23283485
- [Background] Danaher BG, Milgrom J, Seeley JR, Stuart S, Schembri C, Tyler MS, Ericksen J, Lester W, Gemmill AW, Lewinsohn P. Web-Based Intervention for Postpartum Depression: Formative Research and Design of the MomMoodBooster Program. JMIR Res Protoc. 2012 Nov 22;1(2):e18. doi: 10.2196/resprot.2329. PMID 23612274
- [Background] Leung SS, Leung C, Lam TH, Hung SF, Chan R, Yeung T, Miao M, Cheng S, Leung SH, Lau A, Lee DT. Outcome of a postnatal depression screening programme using the Edinburgh Postnatal Depression Scale: a randomized controlled trial. J Public Health (Oxf). 2011 Jun;33(2):292-301. doi: 10.1093/pubmed/fdq075. Epub 2010 Sep 29. PMID 20884642
- [Background] Sword W, Busser D, Ganann R, McMillan T, Swinton M. Women's care-seeking experiences after referral for postpartum depression. Qual Health Res. 2008 Sep;18(9):1161-73. doi: 10.1177/1049732308321736. PMID 18689530
- [Background] Senti J, LeMire SD. Patient satisfaction with birthing center nursing care and factors associated with likelihood to recommend institution. J Nurs Care Qual. 2011 Apr-Jun;26(2):178-85. doi: 10.1097/NCQ.0b013e3181fe93e6. PMID 21372647
- [Background] Dennis CL, McQueen K. The relationship between infant-feeding outcomes and postpartum depression: a qualitative systematic review. Pediatrics. 2009 Apr;123(4):e736-51. doi: 10.1542/peds.2008-1629. PMID 19336362
- [Derived] McCarter DE, Demidenko E, Sisco TS, Hegel MT. Technology-assisted nursing for postpartum support: A randomized controlled trial. J Adv Nurs. 2019 Oct;75(10):2223-2235. doi: 10.1111/jan.14114. Epub 2019 Jul 21. PMID 31222789
- See also: Parenting Stress Index — https://www.apa.org/pi/about/publications/caregivers/practice-settings/assessment/tools/parenting-stress.aspx